CLINICAL TRIAL: NCT00801411
Title: A Randomised Phase 2 Study of Neoadjuvant Docetaxel and Cyclophosphamide Compared to Doxorubicin and Cyclophosphamide in Operable Node Negative Breast Cancer With Normal Topoisomerase IIα Expression
Brief Title: Cyclophosphamide and Docetaxel or Doxorubicin in Treating Women With Newly Diagnosed Breast Cancer That Can Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000624374; SINGAPORE-NCC0705; SANOFI-AVENTIS-NCC0705
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin

ARMS (2):
- Arm I (Experimental): Patients receive cyclophosphamide IV and docetaxel IV over 1 hour on day 1.
  Interventions: Drug: cyclophosphamide; Drug: docetaxel
- Arm II (Active Comparator): Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
Drug: docetaxel — Given IV
  Arms: Arm I
Drug: doxorubicin hydrochloride — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, docetaxel, and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known which chemotherapy regimen is more effective in treating breast cancer.

PURPOSE: This randomized phase II trial is studying cyclophosphamide given together with docetaxel to see how well it works compared with cyclophosphamide given together with doxorubicin in treating women with newly diagnosed breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate tumor pathological complete response rate after neoadjuvant cyclophosphamide in combination with docetaxel vs doxorubicin hydrochloride in women with operable clinically node-negative breast cancer and normal topoisomerase IIα expression.

Secondary

* To assess tumor clinical and pathological overall response rates in patients treated with these regimens.
* To assess the safety and toxicity of these regimens.
* To assess disease-free survival and overall survival of these patients.
* To assess the efficacy of short-course (3 days) filgrastim (G-CSF) as primary and secondary prophylaxis against febrile neutropenia in patients receiving docetaxel and cyclophosphamide.

OUTLINE: This is a multicenter study.

Patients are stratified according to hormone receptor status (estrogen receptor [ER]- or progesterone receptor [PR]-positive vs ER- and PR-negative) and T stage (T2 vs T3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cyclophosphamide IV and docetaxel IV over 1 hour on day 1.
* Arm II: Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1.

In both arms, treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. After completion of neoadjuvant chemotherapy, all patients undergo surgery.

Tumor specimens obtained prior to neoadjuvant chemotherapy are analyzed for topoisomerase IIα gene and protein expression by IHC and FISH. Tissue samples are also collected at surgery for future studies.

After completion of study therapy, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Newly diagnosed disease
  * Operable disease
* Must have clinical T2 (> 2cm) or T3 (> 5 cm) primary tumors with no clinical lymph node involvement (N0)

  * No clinical T4 lesion (e.g., peau d'orange, skin ulceration, satellite nodules, or inflammatory breast cancer)
* No evidence of metastatic disease
* Known hormone receptor status

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status (PS) 0-2 (Karnofsky PS 60-100%)
* Life expectancy > 10 years
* Leukocytes ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal or creatinine clearance ≥ 40 mL/min
* Normal cardiac ejection fraction, defined as ≥ 50% by MUGA scan or 2D-ECHO
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel or other agents used in this study
* No history of pre-existing peripheral neuropathy
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No prior malignancies except curatively treated basal cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No other concurrent investigational or commercial agents or therapies with the intent to treat the patient's malignancy
* No other concurrent chemotherapy, immunotherapy, hormonal cancer therapy, surgery for cancer, or experimental medications
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent antitumor therapy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2008-10

PRIMARY OUTCOMES:
Pathological complete response rate

SECONDARY OUTCOMES:
Clinical and pathological overall response rate
Toxicity as assessed by NCI CTCAE v3.0
Overall survival
Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Wong Nan Soon, MBBS, MRCP, FAMS, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre - Singapore, Singapore